CLINICAL TRIAL: NCT06632938
Title: A Randomized, Single-blind, Placebo-controlled, Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Single Doses of ABBV-382 in Healthy Adult Chinese Volunteers
Brief Title: A Study to Evaluate Adverse Events and How the Drug Moves Through the Body From Subcutaneous (SC) and Intravenous (IV) Doses of ABBV-382 in Healthy Adult Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: M25-081
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-382

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ABBV-382 Dose A (Experimental): Participant will receive a single dose of ABBV-382 Dose A on Day 1 and will be confined to the study site and supervised for approximately 9 days. Participants will be followed-up for approximately 20 weeks.
  Interventions: Drug: ABBV-382
- ABBV-382 Dose A Placebo (Placebo Comparator): Participant will receive a single dose of ABBV-382 Dose A placebo on Day 1 and will be confined to the study site and supervised for approximately 9 days. Participants will be followed-up for approximately 20 weeks.
  Interventions: Drug: Placebo for ABBV-382
- ABBV-382 Dose B (Experimental): Participant will receive a single dose of ABBV-382 Dose B on Day 1 and will be confined to the study site and supervised for approximately 5 days. Participants will be followed-up for approximately 20 weeks.
  Interventions: Drug: ABBV-382
- ABBV-382 Dose B Placebo (Placebo Comparator): Participant will receive a single dose of ABBV-382 Dose B placebo on Day 1 and will be confined to the study site and supervised for approximately 5 days. Participants will be followed-up for approximately 20 weeks.
  Interventions: Drug: Placebo for ABBV-382

INTERVENTIONS:
Drug: ABBV-382 — Subcutaneous (SC) Injection
  Arms: ABBV-382 Dose A
Drug: ABBV-382 — Intravenous (IV) Infusion
  Arms: ABBV-382 Dose B
Drug: Placebo for ABBV-382 — IV Infusion
  Arms: ABBV-382 Dose B Placebo
Drug: Placebo for ABBV-382 — SC Injection
  Arms: ABBV-382 Dose A Placebo

SUMMARY:
The main objectives of this study are to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of single subcutaneous (SC) and intravenous (IV) doses of ABBV-382 in healthy adult Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 27.9 kg/m^2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Females, Non-Childbearing Potential:

  * Premenopausal female with permanent sterility or infertility due to one of following:

    * Permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy)
    * Non-surgical permanent infertility due to Mullerian agenesis, androgen insensitivity, or gonadal dysgenesis OR
  * Postmenopausal, defined as age <= 55 years with no menses for 12 or more months without an alternative medical cause AND a follicle-stimulating hormone (FSH) level >= 30 IU/L.
* Females of Childbearing Potential:

  * If a female does not meet the definition of a female of nonchildbearing potential above, she would be considered a female of childbearing potential.
  * Females of childbearing potential must not be pregnant or breastfeeding.
  * Females of childbearing potential consent to abide by contraception requirements.
  * Females of childbearing potential must agree to avoid pregnancy while taking study drug(s) from Study Day 1 through the end of the study (Day 140) plus an additional 90 days.
  * Females of childbearing potential must use a contraceptive method that is highly effective (with a failure rate of < 1% per year, when used consistently and correctly).
  * Male subjects who are sexually active with a female partner of childbearing potential must agree to use condoms, from Study Day 1 through the end of study (Day 140) plus an additional 90 days, even if the male subject has undergone a successful vasectomy.
  * Male subjects who are not considering fathering a child or donating sperm during the study from Study Day 1 through the end of the study (Day 140) plus an additional 90 days.
* Laboratory values meeting those specified in the protocol.
* A condition of generally good health based on the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).
* In the opinion of the investigator, this participant is a suitable candidate for enrollment in the study.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food, including no history of allergic reaction or anaphylaxis to therapeutic proteins, vaccines, or other parenteral treatments.
* History of hereditary fructose intolerance
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.
* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* Donated blood (including plasmapheresis), lost >= 550 mL blood volume, or received a transfusion of any blood product within 3 months prior to study drug administration.
* Has been previously enrolled in this study.
* Participant has been treated with any investigational drug within 3 months or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.
* Participant has been treated with any anti-α4β7 integrin monoclonal antibody (Ab) or had prior exposure to ABBV-382.
* Participant has received any live vaccine within 4 weeks prior to the first dose of study drug, or expected need of live vaccination during study participation including at least 4 months (120 days) after the last dose of study drug.
* Participant requires any over-the-counter and/or prescription medication, vitamins and/or herbal supplements, with the exception of contraceptives or hormonal replacement therapies for females, on a regular basis.
* Participant uses any medications, vitamins and/or herbal supplements, with the exception of contraceptives or hormonal replacement therapies for females, within the 2-week period prior to study drug administration.
* Receipt of any drug by injection within 30 days or within a period defined by 5 half-lives, whichever is longer, prior to study drug administration, with the exception of parenteral hormonal contraceptives or hormonal replacement therapies for females
* Exposure to antibody-based immunotherapy or previous enrollment in antibody-based immunotherapy clinical trials within a period defined by 5 half-lives prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Approximately Day 140
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of ABBV-382 | Up to Day 112
  Maximum observed serum concentration (Cmax) of ABBV-382.
Time to Cmax (Tmax) of ABBV-382 | Up to Day 112
  Time to Cmax (Tmax) of ABBV-382.
Area Under the Serum Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration (AUCt) of ABBV-382 | Up to Day 112
  Area under the serum concentration-time curve (AUC) from time 0 to the time of last measurable concentration (AUCt) of ABBV-382.
Area Under the Serum Concentration-Time Curve From Time 0 to Infinite Time (AUCinf) of ABBV-382 | Up to Day 112
  AUC from time 0 to infinite time (AUCinf) of ABBV-382.
Terminal Phase Elimination Rate Constant (β) of ABBV-382 | Up to Day 112
  Terminal phase elimination rate constant of ABBV-382.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-382 | Up to Day 112
  Terminal phase elimination half-life of ABBV-382.
Anti-Drug Antibody (ADA) of ABBV-382 | Up to Day 112
  Confirmed Positive ADA Results.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Shanghai Xuhui Central Hospital /ID# 264785, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-081